CLINICAL TRIAL: NCT04797130
Title: The Effect of a Smartphone App With Accelerometer on Patients' Physical Activity: a Randomised Controlled Trial
Brief Title: The Effect of Hospital Fit 2.0 on Patients Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL75126.068.20
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Telemedicine; Internal Medicine; Pulmonary Disease
Keywords: Physical activity; eHealth; Accelerometer; Hospitalization
MeSH Terms: conditions — Lung Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors are blinded for treatment (control group: usual care physiotherapy treatment versus intervention group: usual care physiotherapy treatment and Hospital Fit 2.0 use)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): All subjects eligible for inclusion in this study receive usual care physiotherapy as prescribed by the physician. The number of treatment sessions and content of physiotherapy treatment sessions will depend on the diagnosis and needs of the individual patient. This study will not interfere with the content of the usual care physiotherapy treatment. Patients in the control group will receive an accelerometer, measuring PA, which is applied by the physiotherapist during the first treatment. They receive no other additional intervention. Usual care physiotherapy sessions will take approximately 20-30 minutes per session.
- Intervention group (Experimental): Patients in the intervention group will receive usual care physiotherapy and use Hospital Fit 2.0 (HF) additionally. After the last treatment session (max. 7 days), the therapist will remove the accelerometer and participation in the study will end.
  Interventions: Device: Hospital Fit 2.0

INTERVENTIONS:
Device: Hospital Fit 2.0 — HF consists of a smartphone app combined to an accelerometer. HF provides patients and physiotherapists direct feedback on patients' physical activity behavior.. Individual goals regarding the number of minutes per day spent walking can be set by the therapist. HF also shows patients insight into their own recovery progress. During every treatment, the physiotherapist will evaluate the extent of functional recovery. In addition, Hospital Fit will give physiotherapists the option of creating a patient-specific exercise program supported by videos. During every treatment session, the patient and physiotherapist will evaluate (and if necessary adapt) the amount of activity performed since the previous treatment, the extent of functional recovery and the exercise program.
  Arms: Intervention group

SUMMARY:
The primary objective of this study is to investigate if using Hospital Fit 2.0 as part of the usual care physiotherapy treatment of patients hospitalised at the department of Internal Medicine and the department of Pulmonology in MUMC+ will result in an increase in the amount of PA performed compared to patients who do not use Hospital Fit 2.0 as part of the physiotherapy treatment.

DETAILED DESCRIPTION:
Rationale: Low physical activity (PA) levels are common in hospitalised patients. Digital health tools could be valuable to prevent negative effects of inactivity. We therefore developed Hospital Fit 1.0; a smartphone application with accelerometer, designed for hospitalised patients. It enables objective activity monitoring, provides patients insight in their recovery progress and offers a tailored exercise program. Hospital Fit 1.0 has recently been updated, resulting in the improved Hospital Fit 2.0. Improvements in the accelerometer algorithm are made, a goalsetting and reminder function are added, and data from the app can be linked to the electronic medical record. It is hypothesized that using Hospital Fit 2.0 as part of the physiotherapy treatment of hospitalised patients will result in an increase in the amount of PA performed compared to patients who do not use Hospital Fit 2.0 as part of the physiotherapy treatment.

Objective: To investigate if using Hospital Fit 2.0 as part of the usual care physiotherapy treatment will result in an increase in the amount of PA performed compared to patients who did not use Hospital Fit 2.0 as part of the usual care physiotherapy treatment.

Study design: Assessor blinded randomised controlled trial. Study population: 78 patients hospitalised equally distributed over the department of Internal Medicine and the department of Pulmonology at the Maastricht University Medical Center.

Intervention (if applicable): PA will be measured with an accelerometer until discharge with a maximum of seven days in all patients. The control group receives usual care physiotherapy (n=39), while the intervention group uses Hospital Fit additionally (n=39).

Main study parameters/endpoints: Primary outcome parameter: time spent walking per day (min). Secondary outcome parameters: time spent standing per day (min.), average time spent standing and walking (min.) measured over total measurement time (max. 7 days), number of transitions per day and average number of transitions measured over total measurement time (max. 7 days), number of times walking longer than 5 minutes per day and the average number measured over total measurement time (max.7 days), number of times sitting/lying longer than 30 minutes per day and the average number measured over total measurement time (max. 7 days) and the mILAS score per day (max. 7 days).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden and risks on patients are minimal. The control group will receive usual care physiotherapy and will wear an accelerometer. The intervention group will use Hospital Fit 2.0 additionally. Wearing a small accelerometer and using Hospital Fit 2.0 should not be a burden to patients. The only burden is the time it take to prepare subjects (install app, explain study). No invasive interventions will take place.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years
* Receiving physiotherapy while hospitalised at the department of Internal Medicine department or the department of Pulmonology at the Maastricht University Medical Centre (MUMC+)
* Sufficient understanding of the Dutch language
* Having access to a smartphone
* Able to walk independently 2 weeks before admission, as scored on the Functional Ambulation Categories (FAC >3)

Exclusion Criteria:

* A contraindication to walking (as reported by the attending medical specialists in the medical record)
* A contraindication to wearing an accelerometer, fixed by a hypoallergenic plaster at the upper leg (such as active bilateral upper leg infection, severe edema or bilateral transfemoral amputation)
* Admission at the intensive care department
* Impaired cognition (delirium / dementia) as reported by the attending doctor
* Incapacitated subjects as reported by the attending medical specialist in the medical record. When any doubt arises, the patient will not be considered eligible
* A life expectancy shorter than 3 months as mentioned by the attending medical specialist in the medical record
* Previous participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Time spent walking per day (min.) | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total number of minutes walking per day.

SECONDARY OUTCOMES:
Average time spent walking | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total number of minutes walking divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of seven days
Time spent standing per day (min.) | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total number of minutes walking per day.
Average time spent standing | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total number of minutes standing divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of seven days
Number of transitions from a sedentary position (lying or sitting) to an active position (standing or walking) per day | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total number of transitions from being sedentary (lying or sitting) to being physically active (standing or walking) per day
Average number of transitions from a sedentary position (lying or sitting) to an active position (standing or walking) | Period between inclusion and discharge, with a maximum of seven days
  defined as the total number of transitions divided by the total number of valid measurement days in the period between inclusion and discharge with a maximum of seven days
Number of times walking longer than five minutes | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total number of times per day a patient spent walking for more than 5 minutes continuously without being interrupted by a standing or sedentary activity
Average number of times walking longer than 5 minutes | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total number of times per day a patient spent walking for more than 5 minutes continuously without being interrupted by a standing or sedentary activity, divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of seven days
Number of times sitting/lying longer than 30 minutes | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total numer of times per day a patient spent more than 30 minutes lying and/or sitting without interrupting this behavior with a standing or walking activity.
Average number of times sitting/lying longer than 30 minutes | Period between inclusion and discharge, with a maximum of seven days
  Defined as the total numer of times per day a patient spent more than 30 minutes lying and/or sitting without interrupting this behavior with a standing or walking activity, divided by the total number of valid measurement days in the period between inclusion and discharge, with a maximum of seven days
mILAS score per day | Period between inclusion and discharge, with a maximum of seven days
  Defined as the modified Iowa Level of Assistance Score per day

CONTACTS AND LOCATIONS:
Overall Officials: Antoine F Lenssen, Prof, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
We do not intent to make IPD available to other researchers.